CLINICAL TRIAL: NCT01916044
Title: Evaluation of the Efficiency of the Ultrasound Measure of the Thickness of the Lower Segment Associated With a Rule of Decision to Reduce the Foetal and Maternal Morbidity and Mortality in the Care of the Deliveries of the Women Having a History of Caesarian: a Pragmatic Randomized Trial : Lustrial
Brief Title: Ultrasound Measure of the Thickness of the Lower Segment in Women Having a History of Caesarian
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P111103
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Lower Uterine Segment; Labor
Keywords: caesarean,; trial of labor,; ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lower Uterine Segment Ultrasound (Experimental): Measure of Uterine Segment by Ultrasound
  Interventions: Other: Ultrasound
- control (No Intervention): no measure of Uterine Segment Ultrasound

INTERVENTIONS:
Other: Ultrasound — Measure of Uterine Segment by Ultrasound
  Arms: Lower Uterine Segment Ultrasound

SUMMARY:
The rate of caesarians dramatically increased for 15 years. The main indication of caesarian became the iterative caesarian of principle because of a history of caesarian. Any attempt of reduction of the rate of caesarians should thus focus on the indications of iterative principal caesarean. Nevertheless, the main reason usually evoked to justify a reduction of the attempts of low way after caesarian is the concern generated by the risk of uterine break during the trial of labor. Yet, there is no reliable method to predict this risk of uterine break. A way of interesting research consists in estimating the potential profits of the echography of the scar lower segment. Indeed, the echography can be useful to determine the specific risk of uterine break of a patient by measuring the thickness of the lower segment of the womb.

The strong negative predictive value of the echography of the lower segment on the risk of uterine break should encourage the women encircled to accept a trial of labor. That is why, this examination associated with a rule of decision could help to decrease the rate of iterative elective caesarians and especially to decrease the mortality and the foetal and maternal morbidity connected to the trial of labor among the patients having a history of caesarian.

DETAILED DESCRIPTION:
"Lower Uterine Segment Trial (LUSTrial)" Evaluation of the efficiency of the ultrasound measure of the thickness of the lower segment associated with a rule of decision to reduce the foetal and maternal morbidity and mortality in the coverage of the deliveries of the women having a history of caesarian: a pragmatic randomized trial

Aim Evaluation of the efficiency of the ultrasound measure of the thickness of the lower segment associated with a rule of decision to reduce the foetal and maternal morbidity and mortality in the coverage of the deliveries of the women having a history of caesarian Methodology Randomized trial, multicentric, open, in two parallel arms.

Evaluated treatments:

Between 36+0 and 38+6 weeks of amenorrhea, the patients will be invited to participate in the study. After agreement, the patients respecting the criteria of inclusion and not inclusion will be randomized in two groups:

GROUP A (experimental group) : The ultra sound measure of the thickness of the lower segment will be realized in a way standardized by expert sonographers. The patient will be informed that in case of measure:

* superior at the threshold of 3.5 mm, her will be considered " a low risk " by complications and will be encouraged to try a event of the work
* subordinate or equal at the threshold of 3.5 mm, her will be considered " at risk " by complications and will be encouraged to give birth by iterative elective caesarian.

GROUP B (control group) : The ultra sound measure of the lower segment will not be realized. The mode of delivery will be decided according to the current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* unique pregnancy
* gestational age between 36 SA and 38SA +6 days
* cephalic presentation
* lower uterine segment section's history
* sign consent

Exclusion Criteria:

* age < 18 years
* history of longitudinal incision's caesarean
* iterative caesarean indication
* multiple pregnancy
* placenta praevia
* patient refuse trial of labor
* absent consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2955 (Actual)
Dates: Start 2013-07-11; Primary Completion 2018-05-11 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Composite criterion including maternal and neonatal parameters | at 3 days post partum
  rupture uterine, uterine dehiscence, hysterectomy, deep venous thromboembolic complications, transfusion, endometritis, maternal mortality, foetal mortality antepartum, intrapartum foetal mortality, ischemic hypoxic encephalopathy, neonatal mortality

SECONDARY OUTCOMES:
Uterine rupture | at 3 days post partum
Uterine dehiscence | at 3 days post partum
  Maternal morbidity
Antepartum and intrapartum mortality | 3 days post partum
  Foetal mortality
Hypoxic-ischemic encephalopathy | at 3 days post partum
  New born morbidity
Thromboembolic complications | at 3 days post partum
  Maternal morbidity
Hysterectomy | at 3 days post partum
  Maternal morbidity
Transfusion | at 3 days post partum
  Maternal morbidity
Endometritis | at 3 days post partum
  Maternal morbidity
Rate of elective caesarean sections and of caesarean sections during labor | at 1 day post partum
Perineal tears of the 3rd and 4th degree | at 1 day post partum

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Rozenberg, MD, PhD, Principal Investigator — CHI Poissy
Locations (1):
- CHI Poissy Saint Germain, Poissy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rozenberg P, Senat MV, Deruelle P, Winer N, Simon E, Ville Y, Kayem G, Porcher R, Perrodeau E, Desbriere R, Boutron I; Groupe de Recherche en Obstetrique et Gynecologie. Evaluation of the usefulness of ultrasound measurement of the lower uterine segment before delivery of women with a prior cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2022 Feb;226(2):253.e1-253.e9. doi: 10.1016/j.ajog.2021.08.005. Epub 2021 Aug 9. PMID 34384777
- [Derived] Rozenberg P, Deruelle P, Senat MV, Desbriere R, Winer N, Simon E, Ville Y, Kayem G, Boutron I; Groupe de recherche en obstetrique et gynecologie. [Lower Uterine Segment Trial: A pragmatic open multicenter randomized trial]. Gynecol Obstet Fertil Senol. 2018 Apr;46(4):427-432. doi: 10.1016/j.gofs.2018.03.005. Epub 2018 Apr 4. French. PMID 29625873